CLINICAL TRIAL: NCT05644548
Title: Retinal Vascular Manifestations in Patients With Common Internal Diseases on Optical Coherence Tomography Angiography
Brief Title: Retinal Vascular Manifestations in Patients With Common Internal Diseases on OCTA Tomography Angiography
Status: Recruiting | Type: Observational
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: YuHe2022
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Hypertension; Diabetes Mellitus; Dyslipidemias
Keywords: OCTA; Hypertension; Diabetes; Dyslipidemias
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Hypertension: No intervention
  Interventions: Other: No intervention
- Diabetes mellitus: No intervention
  Interventions: Other: No intervention
- Dyslipidemia: No intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Hypertension, diabetes mellitus, and dyslipidemia are common internal diseases, and all diseases are atherosclerosis risk factors. Previous studies applied color fundus photography to analyze retinal vascular changes (including exudation, hemorrhage, neovascularization, etc.) in patients with hypertension or diabetes, but the examination results could not be quantified.

This study intends to apply optical coherence tomography angiography (OCTA) to examine retinal vessels. This method has the following advantages: 1) It can quantify vascular changes, and 2) It is noninvasive and reproducible for patients' follow-up.

This study was designed to investigate retinal vascular changes in patients with hypertension, diabetes, and dyslipidemia on OCTA. We will collect the patients' general information (gender, age), comorbidities, medications, blood lipids, blood glucose, carotid ultrasound, ankle-brachial index, ambulatory blood pressure monitoring, color fundus photography, and OCTA results. We will follow up with the patients for five years and conduct the mentioned examinations once a year. We will also investigate the correlation between systemic atherosclerosis (such as coronary artery stenosis, and carotid artery stenosis) and retinal vasculopathy in patients with these diseases.

DETAILED DESCRIPTION:
Patients with hypertension, diabetes mellitus, or dyslipidemia, who go to the department of geriatric medicine, Beijing Tongren Hospital from March 2022 to December 2023 will be included. We will collect general information, comorbidities, medication, laboratory tests, and examination results. These patients will be followed up for 5 years with a yearly collection of comorbidities, medication, laboratory tests, and examination results.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypertension
* Or patients with diabetes
* Or patients with dyslipidemia
* Agree to participate in this study

Exclusion Criteria:

* Patients with malignant tumors
* Patients with autoimmune diseases
* Patients with immunodeficiency disease
* Disagree to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the geriatric department of Beijing Tongren Hospital, China. Beijing Tongren Hospital is a third-class hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Vascular density of the retina | up to 5 years of follow-up.
  percent

SECONDARY OUTCOMES:
the foveal avascular zone (FAZ) size of the retina | When participating in the study, and once a year during 5 years of follow-up.
  mm2

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma JB, Qin MZ, Cao K, Zhang YP, Guo CX. Control of blood pressure and blood glucose levels has important clinical significance to the retina. BMC Ophthalmol. 2025 Jul 1;25(1):368. doi: 10.1186/s12886-025-04164-y. PMID 40597972
- [Derived] He Y, Qin MZ, Cao K, Zhang YP, Jiao X, Zhang Z, Wang GH, Liu Q, Liu Q, Ma JB, Jiang X, Guo CX. Assessment of the impact of low-density lipoprotein cholesterol on retinal vessels using optical coherence tomography angiography. Lipids Health Dis. 2024 Sep 16;23(1):301. doi: 10.1186/s12944-024-02287-7. PMID 39285295